CLINICAL TRIAL: NCT01983956
Title: A Structured Early Palliative Care Intervention for Patients With Advanced Cancer - a Randomized Controlled Trial With a Nested Qualitative Study (SENS Trial)
Acronym: SENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 102/13; 2401 (Other: Direktion Lehre und Forschung, Inselspital (study number)); 406740_145088/1 (Other Grant/Funding Number: Schweizerischer Nationalfonds)
Record Dates: First submitted 2013-11-05; First posted 2013-11-14 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Advanced Cancer
Keywords: early palliative care; patient empowerment; cancer; assessment; end of life
MeSH Terms: conditions — Patient Participation; Neoplasms; Death

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): The structured approach intervention with the SENS model is based on the bio-psycho-social-spiritual model of care and the WHO definitions of palliative care as well as the NCCN Practice Guidelines for Palliative Care. It supports the assessment of areas and complexity of concerns from the patient perspective, determines the priority and structures the support needed. The intervention is performed by palliative care physicians and nurses collaboratively. It is utilized as baseline assessment and afterwards integrated in each routine oncology care out-patient and in-patient visit. Depending on the goals it may be applied between routine visits. In addition, patients will receive usual oncology care throughout the study period.
  Interventions: Behavioral: SENS model
- Control arm (No Intervention): Patients in the usual care group will receive routine oncology care throughout the study. This incorporates a routine assessment according to the standard SAKK - protocol which assesses overall symptoms. Patients are not seen by nurses during a routine visit to the outpatient clinic unless they need a blood withdrawal or any intravenous or subcutaneous treatment. Only nursing staff of the palliative care unit is familiar with using the SENS-assessment instrument. Participants assigned to usual care may meet with the palliative care service on request according to established practice.

INTERVENTIONS:
Behavioral: SENS model — Palliative care with a structured approach (SENS model) based on the bio-psycho-social-spiritual model of care, the WHO definitions of palliative care as well as the National Comprehensive Cancer Networks (NCCN) Practice Guidelines for Palliative Care. The approach supports the assessment of areas and complexity of concerns from the patient perspective, determines the priority and structures the support needed. The intervention is performed by palliative care physicians and nurses collaboratively. It is utilized as baseline assessment and afterwards integrated in each routine oncology care out-patient and in-patient visit. Depending on the goals it may be applied between routine visits. In addition, patients will receive usual oncology care throughout the study period.
  Arms: Experimental arm

SUMMARY:
It is assumed that an early palliative care structured by SENS (a systematic, problem-based assessment system) in addition to standard oncology care compared with standard oncology care alone relieves distress in patients with advanced cancer at the end of life.

The primary objective of the trial is to determine the effectiveness of early palliative care intervention, structured by SENS (a systematic, problem-based assessment system) in addition to standard oncology care, compared with standard oncology care alone to relieve distress a) in patients with advanced cancer until death, and b) in caregivers. The secondary objectives are to determine whether the introduction of SENS improves quality of life, prolongs overall survival, ameliorates distress of caregivers, reduces health care costs and medical resource utilization (less aggressive treatment in the last weeks of life).

DETAILED DESCRIPTION:
Background

Intervention (performed by specialist palliative care teams): The structured approach intervention is based on NCCN Practice Guidelines for Palliative Care, part of Gold Standard Framework (GSF) and the WHO definition of Palliative Care. It supports the assessment of areas and complexity of concerns from the patient perspective, determining priorities and structures the support needed. SENS stands for: Symptom-management, instruction for self administration of medication etc. End of life decision-making: explicit definition of own goals and priorities; Network organization including anticipatory planning of emergency situations

Support of the carers: implementation of support systems for the caring family members

The standardized intervention (based on prepared educational tool kit including a patient prompt sheet) is performed by a palliative care physician and nurse collaboratively after randomization and consent. The intervention is undertaken only once (after baseline questionnaire and before first follow-up questionnaire). There is a total of 4 questionnaires in the first 6 months. In addition, patients will receive usual oncology care throughout the study period (see below).

Usual Oncology care (performed by oncological out- and inpatient clinics): Usual care incorporates a routine assessment according to national protocols, which assesses overall symptoms and current complaints from other domains. Participants assigned to usual care may meet with the palliative care service on request according to established practice but without following the SENS approach (subgroup analysis will be performed).

Main eligibility criteria

Patients >/= 18 years of age who signed informed consent with understanding of the study procedures and the investigational nature of the study with one of the following cancer types:

* Diagnosed within the last 16 weeks
* Metastatic or locally advanced, not amenable to curative treatment, non- small cell lung cancer (NSCLC), or
* Metastatic or locally advanced, not amenable to curative treatment, colorectal cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, prostate cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, breast cancer with visceral and/or brain metastasis, or
* Metastatic or locally advanced, not amenable to curative treatment, bladder/ urothelium cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, pancreatic cancer
* Diagnosis is histologically confirmed
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2

Exclusion criteria

* Presence of delirium or dementia or other reason for lack of ability to give informed consent
* Inability to communicate adequately in German
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly
* Patients already receiving care from an inpatient palliative care service

Outcomes Primary outcomes

* Distress over six month as measured with the National Comprehensive Cancer Network (NCCN) Distress thermometer Secondary outcomes
* Quality of life as measured by Functional Assessment of Cancer Therapy - General (FACT-G)
* Palliative Outcome Scale (POS)
* Overall survival
* Location of death
* Health care utilization

Objective

The primary objective of the trial is to determine the effectiveness of early palliative care structured by SENS (a systematic, problem-based assessment system) in addition to standard oncology care compared with standard oncology care alone to relieve distress in patients with advanced cancer at the end of life.

The secondary objectives are to determine whether the introduction of SENS improves quality of life and prolongs overall survival in these patients, reduces health care costs and medical resource utilization.

The primary objective of the nested qualitative study is to identify characteristics and reasons for the added value as well as failure of a compulsory problem-based assessment system (SENS) in advanced cancer patients.

Methods

Design Multicenter, two-arm, parallel-group, randomized-controlled trial with a nested qualitative study (content analysis)

Experimental arm:

Palliative care with a structured approach (SENS model) based on the bio-psycho-social-spiritual model of care. The approach supports the assessment of areas and complexity of concerns from the patient perspective, determines the priority and structures the support needed. The intervention is performed by palliative care physicians and nurses collaboratively.

Control arm: Patients in the usual care group will receive routine oncology care throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed within the last 16 weeks
* Metastatic or locally advanced, not amenable to curative treatment, non- small cell lung cancer (NSCLC), or
* Metastatic or locally advanced, not amenable to curative treatment, colorectal cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, prostate cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, breast cancer with visceral and/or brain metastasis, or
* Metastatic or locally advanced, not amenable to curative treatment, bladder/ urothelium cancer, or
* Metastatic or locally advanced, not amenable to curative treatment, pancreatic cancer
* Diagnosis is histologically confirmed
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2
* At least 18 years of age at the time of enrolment
* Signed informed consent with understanding of the study procedures and the investigational nature of the study

Exclusion Criteria

* Presence of delirium or dementia or other reason for lack of ability to give informed consent
* Inability to communicate adequately in German
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly
* Patients already receiving care from an inpatient palliative care service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2020-04-25 (Estimated)

PRIMARY OUTCOMES:
Distress over six month as measured with the National Comprehensive Cancer Network (NCCN) Distress thermometer | Six months

SECONDARY OUTCOMES:
Quality of life as measured by Functional Assessment of Cancer Therapy - General (FACT-G) | Six months
Palliative Outcome Scale (POS) | Six months
Overall survival | four years
Location of death | Six months
Health care utilization | Six months
  Measured using the questionnaire of Stanford Patient Education Research Centre.

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Eychmüller, Prof. Dr. med., Principal Investigator — University Hospital Berne; University Center for Palliative Care
Locations (3):
- Switzerland (3):
  - Dep. of Haematology, Oncology, Infectiolog, Laboratory Medicine and Spital-pharmacy (DOLS); University Center for Palliative Care, Bern University Hospital, 3010 Bern, Bern
  - Kantonsspital Luzern, Medizinische Onkologie, Schwerpunktabteilung Palliative Care, Lucerne
  - Kantonsspital St. Gallen, Palliativzentrum, Sankt Gallen

REFERENCES:
- [Background] Abstracts of the ninth annual meeting of the Japanese Society of Biorheology. Ehime, Japan, 13-15 June 1986. Biorheology. 1986;23(5):513-47. doi: 10.3233/bir-1986-23507. No abstract available. PMID 3651574
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Zhang B, Wright AA, Huskamp HA, Nilsson ME, Maciejewski ML, Earle CC, Block SD, Maciejewski PK, Prigerson HG. Health care costs in the last week of life: associations with end-of-life conversations. Arch Intern Med. 2009 Mar 9;169(5):480-8. doi: 10.1001/archinternmed.2008.587. PMID 19273778
- [Background] Zmorski T, Fischer-Cornelssen KA. [Clinical experiences with the new-generation anxiolytic agent cloxazolam--a double-blind study]. Schweiz Rundsch Med Prax. 1985 Jul 2;74(27):728-34. No abstract available. German. PMID 2862687
- [Background] Hawkes AL, Hughes KL, Hutchison SD, Chambers SK. Feasibility of brief psychological distress screening by a community-based telephone helpline for cancer patients and carers. BMC Cancer. 2010 Jan 12;10:14. doi: 10.1186/1471-2407-10-14. PMID 20067645
- [Derived] Maessen M, Fliedner MC, Gahl B, Maier M, Aebersold DM, Zwahlen S, Eychmuller S. An economic evaluation of an early palliative care intervention among patients with advanced cancer. Swiss Med Wkly. 2024 Feb 16;154:3591. doi: 10.57187/s.3591. PMID 38579309
- [Derived] Eychmuller S, Zwahlen S, Fliedner MC, Juni P, Aebersold DM, Aujesky D, Fey MF, Maessen M, Trelle S. Single early palliative care intervention added to usual oncology care for patients with advanced cancer: A randomized controlled trial (SENS Trial). Palliat Med. 2021 Jun;35(6):1108-1117. doi: 10.1177/02692163211005340. Epub 2021 Apr 28. PMID 33908288
- [Derived] Fliedner M, Zambrano S, Schols JM, Bakitas M, Lohrmann C, Halfens RJ, Eychmuller S. An early palliative care intervention can be confronting but reassuring: A qualitative study on the experiences of patients with advanced cancer. Palliat Med. 2019 Jul;33(7):783-792. doi: 10.1177/0269216319847884. Epub 2019 May 9. PMID 31068119